CLINICAL TRIAL: NCT02107131
Title: Evaluation of ReAding Speed, Contrast Sensitivity, and Work Productivity in Working Individuals With Diabetic Macular Edema Following Treatment With Intravitreal Ranibizumab
Brief Title: Performance Assessment Tests in Working Individuals With DME Following Treatment With Ranibizumab
Acronym: ERASER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29184s
Record Dates: First submitted 2014-04-02; First posted 2014-04-08 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monthly Intravitreal ranibizumab 0.3mg (Active Comparator): Monthly Intravitreal ranibizumab 0.3mg injections.
  Interventions: Drug: Intravitreal ranibizumab 0.3mg
- PRN Intravitreal ranibizumab 0.3mg (Active Comparator): PRN Intravitreal ranibizumab 0.3mg injections.
  Interventions: Drug: Intravitreal ranibizumab 0.3mg

INTERVENTIONS:
Drug: Intravitreal ranibizumab 0.3mg

SUMMARY:
Performance assessment testing may be a useful tool to evaluate the impact of ranibizumab on day-to-day visual function in patients with Diabetic Macular Edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 18 ≤ x ≤ 65 years and currently employed at the baseline study visit
* Diagnosis of diabetes mellitus (type 1 or 2)

  o Any one of the following will be considered to be sufficient evidence that diabetes is present:
* Current regular use of insulin for treatment of diabetes
* Current regular use of oral anti-hyperglycemia agent for the treatment of diabetes
* Clinical evidence of retinal thickening due to macular edema involving the center of the macula, associated with diabetic retinopathy.
* Central diabetic macular edema present on clinical examination or or evidence indicating disease activity on spectral domain OCT.
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
* Participation in another ocular investigation or trial simultaneously
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110)
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse)
* Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema
* An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis or geographic atrophy)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gas)
* Evidence of active neovascularization of the iris or retina
* Evidence of central atrophy or fibrosis in the study eye
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* Previous use of intraocular or periocular corticosteroids in the study eye in the previous 120 days
* Previous treatment with anti-angiogenic drugs in the study eye i.e. pegaptanib sodium, bevacizumab, ranibizumab, aflibercept within 120 days prior to baseline
* History of vitreous surgery in the study eye
* History of cataract surgery within 3 months of enrollment.
* History of YAG capsulotomy within 2 months of enrollment.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled glaucoma (pressure >30) despite treatment with glaucoma medications.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gordon, PhD, Study Director — California Retina Consultants
Locations (6):
- United States (6):
  - California Retina Consultants - Bakersfield, Bakersfield, California
  - California Retina Consultants, Oxnard, California
  - California Retina Consultants, Palmdale, California
  - California Retina Consultants - Santa Barbara Office, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - California Retina Consultants, Visalia, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Monthly: Monthly Intravitreal ranibizumab 0.3mg
- PRN Group: PRN Intravitreal ranibizumab 0.3mg
Period: Overall Study
Arm/Group | Monthly | PRN Group
Started | 20 | 20
Completed | 12 | 11
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 4 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — mental instability | 1 | 0
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly | PRN Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: A Change Between Two Time Points is Reported for Maximum Reading Speed
Description: A change between two time points (Baseline and 12 months) is reported for Maximum Reading Speed.
Time Frame: Month 12
Population: MNREAD words per minute
Measure: Mean (Standard Deviation); unit: words per minute
Arm/Group | Monthly | PRN Group
Number analyzed (Participants) | 12 | 11
words per minute | 161.94 (43.56) | 167.65 (32.30)

2. Secondary Outcome: Change in Activity Productivity
Description: To evaluate the mean change in activity impairment from baseline to 12 months using and activity impairment questionnaire. Scale is from 0-10 with 0 being lowest (no effect on my daily activities) and 10 being highest (completely prevented me from doing my daily activities).
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Monthly | PRN Group
Number analyzed (Participants) | 12 | 9
Units on a scale | -2.25 (3.14) | -0.78 (2.44)

3. Secondary Outcome: Change in Visual Acuity
Description: To determine the mean change in best-corrected visual acuity on ETDRS visual acuity chart at a starting distance of 4 meters from baseline. Visual function of the study eye was assessed using the ETDRS protocol, which is a widely accepted international standard. A higher letter score represents better functioning.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Monthly Intravitreal Ranibizumab 0.3mg: Monthly Intravitreal ranibizumab 0.3mg injections.
  Intravitreal ranibizumab 0.3mg
- PRN Intravitreal Ranibizumab 0.3mg: PRN Intravitreal ranibizumab 0.3mg injections.
  Intravitreal ranibizumab 0.3mg
Arm/Group | Monthly Intravitreal Ranibizumab 0.3mg | PRN Intravitreal Ranibizumab 0.3mg
Number analyzed (Participants) | 12 | 12
Letters | 17.42 (15.13) | 14.92 (11.60)

4. Secondary Outcome: Change in Contrast Sensitivity
Description: To measure the mean change in contrast sensitivity scores on Pelli-Robson charts from baseline. Scale in assessing the log of the contract sensitivity score (CS score) is from 0-2.25, with 0 being no letters read on the contrast sensitivity chart, and 2.25 being all letters read on the contrast sensitivity chart. Total CS score = [(total # letters correct - 3) x 0.05].
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Monthly | PRN Group
Number analyzed (Participants) | 11 | 11
Units on a scale | 0.39 (0.45) | 0.26 (0.40)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Arm/Group | Monthly | PRN Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 5/20 | 4/20
Other Adverse Events (participants affected / at risk) | 15/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monthly (N=20) | PRN Group (N=20)
Myocardial infarction (Cardiac disorders) | 1 | 1
fractured humerus and tibia (Injury, poisoning and procedural complications) | 1 | 0
Septic Knee (Infections and infestations) | 1 | 0
stress, cardiomyopathy, acute renal disfunction (Cardiac disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
lower back and abdominal pain (Gastrointestinal disorders) | 1 | 0
congestive heart failure (Cardiac disorders) | 1 | 0
Urinary Tract Infection with Sepsis (Renal and urinary disorders) | 0 | 1
Blurry Vision (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monthly (N=20) | PRN Group (N=20)
Upper respiratory infection (Reproductive system and breast disorders) | 2 | 4
Flu/cold (Infections and infestations) | 8 | 2
Eye Pain (Eye disorders) | 3 | 4
Eye redness (Eye disorders) | 4 | 5
Eye Itchiness (ocular pruitis) (Eye disorders) | 3 | 0
Blurry/distorted vision (Eye disorders) | 1 | 2
Allergies/ Congestion (Immune system disorders) | 2 | 0
Shingles (Infections and infestations) | 0 | 1
Floaters (Eye disorders) | 3 | 1
Photophobia (Eye disorders) | 1 | 1
Selective Laser Trabeculotomy (Surgical and medical procedures) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Anxiety (General disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
fall (General disorders) | 1 | 1
diarrhea (Gastrointestinal disorders) | 2 | 0
leg injury (Injury, poisoning and procedural complications) | 2 | 1
herniea/hernia repair (Surgical and medical procedures) | 1 | 0
Cataract Extraction (Surgical and medical procedures) | 1 | 0
Subconjunctival Hemorrhage (Eye disorders) | 2 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Heart Infection (Infections and infestations) | 1 | 1
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Hospitalization for swelling and fluid (General disorders) | 1 | 0
Kidney stone (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02107131/Prot_SAP_000.pdf